CLINICAL TRIAL: NCT06403735
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of QLC1101 Monotherapy in the Treatment of Patients With Advanced Solid Tumors Harboring a KRAS G12D Mutation
Brief Title: A Phase I Clinical Study of QLC1101 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLC1101-101
Record Dates: First submitted 2024-04-10; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Non-small Cell Lung Cancer; Colorectal Cancer; Pancreatic Cancer; Solid Tumor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QLC1101 (Experimental): patients with advanced solid tumors harboring a KRAS G12D mutation were administrated with QLC1101 orally in a total of 6 dose groups at 100,200,400,600,900, and 1200 mg BID
  Interventions: Drug: QLC1101

INTERVENTIONS:
Drug: QLC1101 — QLC1101 is an innovative small molecule inhibitor targeting KRAS G12D with independent intellectual property rights developed by Qilu Pharmaceutical Co., Ltd.QLC1101 can prevent GTP/GDP nucleotide exchange and/or the formation of KRAS G12D/GTP/RAF1 complex and inhibit mutant KRAS-dependent signal transduction by specifically binding to the KRAS G12D target, thereby inhibiting the generation of KRAS G12D mutant tumors.

SUMMARY:
QLC1101 is a selective reversible inhibitor of KRAS G12D, with the dosage form of capsules and administration route of oral administration. In the first-in-humans (FIH) study, the sponsor will explore the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of QLC1101 in subjects with advanced solid tumors harboring a KRAS G12D mutation. The FIH study includes dose escalation, PK expansion, and efficacy expansion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed advanced (metastatic or unresectable) solid tumors harboring a KRAS G12D mutation. Sign the ICF.
2. Those who fail or are unable to tolerate standard treatment, lack standard treatment, or refuse to receive standard treatment;
3. Those who are able to swallow and retain oral medication and must not have any clinically significant gastrointestinal abnormality that may alter absorption;
4. Subjects who have at least one measurable lesion documented by computed tomography (CT) and/or magnetic resonance imaging (MRI) as confirmed by the investigator per the RECIST v1.1 criteria.
5. ECOG PS score: 0 or 1;
6. Expected survival time ≥ 3 months;
7. Adequate organ function at screening:

Exclusion Criteria:

1. Previously treated with inhibitors against KRAS G12D mutation;
2. The period of time prior to the first dose of investigational product should be at least 28 days from previous treatment or at least 5 half-lives
3. Known immediate or delayed hypersensitivity or idiosyncratic reaction to the ingredients of the preparation used in the trial;
4. Presence of other active malignant tumors in addition to primary tumors;
5. Presence of serious lung diseases at screening;
6. Clinically significant gastrointestinal disorders or other conditions that seriously interfere with drug absorption;
7. Severe hereditary or acquired hemorrhagic diathesis or coagulation disorders;
8. Complicated with clinically significant cardiovascular and cerebrovascular disorders;
9. History of allogeneic hematopoietic stem cell transplantation or organ transplantation (except corneal transplantation);
10. Presence of known mental disorders, epilepsy, dementia, or alcohol and drug abuse that may affect the compliance with study requirements;
11. the investigator determines that participation in the study is not in the best interest of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 25 days after the first dose
  Subjects in this phase will be treated with single oral administration of QLC1101, observed for 4 days, and if tolerant, treated with repeated oral administration of QLC1101 twice daily for 21 consecutive days. After completing the DLT observation (the 25 days after the first dose as the DLT observation period), the subject will continue to receive repeated-dose treatment of Cycle 2 and subsequent cycles.
MTD (or MAD) | 1 year
  the maximum tolerated dose (MTD) or maximum administered dose (MAD, if MTD fails to be determined) of QLC1101 monotherapy
RP2D | 1.5 years
  the recommended phase II dose of QLC1101 monotherapy

SECONDARY OUTCOMES:
Preliminary efficacy endpoints | 3 years
  Objective response rate (ORR)
Preliminary efficacy endpoints | 3 years
  overall survival (OS)

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - Harbin Medical university cancer hospital, Harbin, Heilongjiang
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Shanghai east hospital, Shanghai, Shanghai Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan